CLINICAL TRIAL: NCT03309631
Title: Clinical Validation of ThyroidPrint: A Gene Expression Signature for Diagnosis of Indeterminate Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Geneprodx (Unknown)
Responsible Party: Principal Investigator, Hernán González, Associate Professor, Pontificia Universidad Catolica de Chile
Other Study IDs: GPDX-001
Record Dates: First submitted 2017-10-01; First posted 2017-10-13 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Indeterminate Thyroid Cytology
Keywords: Gene classifier

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fine needle Aspiration of a thyroid nodule
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: In vitro Diagnostic

SUMMARY:
A clinical trial is proposed, to clinically validate, in a US population, the diagnostic performance of a new genetic test (ThyroidPrint). It will determine the nature of thyroid nodules that have been informed as indeterminate by cytology through a fine needle aspiration (FNA). The Genetic Classifier for Indeterminate Thyroid Nodules is a test that determines the expression of a panel of 10 biomarkers (CXCR3, CCR3, CXCl10, CK19, TIMP1, CLDN1, CAR, XB130, HO-1 and CCR7). Gene expression data is analyzed through an algorithm that generates a composite score that predicts the risk of malignancy. It´s intended use is for patients with thyroid cytology as indeterminate (Bethesda III and IV, according to The Bethesda System for Reporting Thyroid Cytopathology). This test uses a fine needle aspiration (FNA) sample.

DETAILED DESCRIPTION:
Thyroid nodules are a very frequent condition reaching up to 30-40% of the adult population. Although most thyroid nodules have little clinical significance, in many cases a fine needle aspirate (FNA) biopsy will be performed to determine its nature. In 70% of cases, a FNA will be reported as benign and in 10% of cases as cancer. However, the remaining 20% of cases the thyroid nodule will be reported as indeterminate. The latter patients have a risk of malignancy ranging from 15 to 25%, and in most cases the patient will undergo thyroid lobectomy or total thyroidectomy to determine the final pathology, resulting in an unacceptable number of unnecessary surgeries. This has a major health impact, including surgical risks and permanent hormonal supplementation, as well as unwarranted health costs estimated at 1.6 billion USD. Therefore, there is a need for diagnostic tools in order to improve the diagnostic accuracy of the FNA and avoidance of the high rate of unnecessary surgeries.

GeneproDx has developed a gene expression signature to improve the diagnostic accuracy of FNA biopsy of thyroid nodules reported as indeterminate. The ThyroidPrint diagnostic measures the expression of 10 genes in a FNA sample. It combines the results of the 10 biomarkers using a proprietary algorithm to predict benign thyroid nodules. This assay is classified as multi-analyte algorithm assays (MAAA).

The biomarkers consist of multiplex TaqMan® gene expression assays run on Qiagen's Rotor-Gene Q MDx RT-PCR IVD Platform instrument, which is a FDA cleared instrument. The following 10 genes comprise the biomarker panel: CXCR3, CCR3, CXCL10, CK19, TIMP1, CLDN1, CAR, XB130, HO-1 and CCR7. Each gene run in a multiplex configuration with two reference genes. Each assay is performed with Research Use Only (RUO) kits and reagents on a FDA cleared instrument.

ThyroidPrint has been developed using two different cohorts of samples, a training set and a testing set. Using linear discriminant analysis, the training set identified the final biomarker panel including; CXCR3, CCR3, CXCL10, CK19, TIMP1, CLDN1, CAR, XB130, HO-1 and CCR7. In brief, the biomarkers have the following significance. CCR3 and CCR7 are chemokine receptors that are highly expressed in papillary thyroid cancer tumor cells. CXCR3 is also a chemokine receptor and along with its receptor, CXCL10, are detected in thyroid autoimmune disease. CAR is a G-couple receptor and has been shown to be involved in cancer and has decreased expression in parathyroid adenoma. CK19 is a keratin and has been used in thyroid tumors to recognize papillary carcinomas. CLDN1 is a structural protein and has been shown to be differentially expressed in tumors compared to normal tissue and has increased mRNA levels in papillary thyroid carcinoma. XB130 is also a structural protein and its expression has been demonstrated in papillary thyroid carcinoma. TIMP1 is a protease inhibitor with mRNA levels increased in advanced stages of thyroid carcinoma. HO- 1 is an oxygenase and its expression has correlates with tumor aggressiveness in thyroid cancer. In the final classifier, the expression of each gene was ̈weighted ̈ based on its individual relative classifying ability. The cutoff score was chosen in the ROC curve generated in the training set based on a minimum Sensitivity of 92% to guarantee a high Negative Predictive Value (>95%). This cutoff score offered a Specificity of 83%.An independent testing set of samples reproduced the diagnostic performance observed in the training set and showed consistent results in FNA samples. The assay has proven to accurately predict benign nodules in thyroid FNA samples with a Negative Predictive Value of 96% and Specificity of 83% in both cohorts. The definitive validation of an MAAA requires a final validation set, which analyzes samples that will be used in the routine clinical setting; in this case indeterminate thyroid nodules samples. In addition, in order to show clinical validity, the validation set must be performed, as a statistically powered multi-institutional trial to assure that the data is applicable to a broad population spectrum and has appropriate confidence intervals. A first, statistically powered, multi-institutional trial is currently underway in Chile to prove Clinical Validity. This trial includes 8 sites and will recruit approximately 3000 FNA to be completed by December 2017.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing FNA of a thyroid nodule.
2. Thyroid nodule greater 1cm
3. Age greater 18 years old.

Exclusion Criteria:

1. Thyroid nodule greater 1cm
2. Patients less than 18 years old,
3. Previous history of coagulation disorders and patients.
4. Ultrasound evidence of malignant cervical adenopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a thyroid nodule recommended to undergo a fine needle aspiration (FNA) cytology evaluation by there attending physician are invited to participate in the trial. At the time of the FNA an additional sample will be collected for molecular testing. Only patients with an indeterminate result (Bethesda III and IV) will continue in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Ability to predict Benign thyroid nodules. | 24 months
  This will be determined by the Negative Predictive Value
Ability to predict Malignant thyroid nodules. | 24 months
  This will be determined by the Positive Predictive Value
Sensitivity of the test | 24 months
  Number of true positives cases
Specificity of the test | 24 months
  Number of true negative cases

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zafareo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - Avantt Research, Guntersville, Alabama
  - Stanford University, Palo Alto, California
  - Lee Moffit Cancer Center, Tampa, Florida
  - Tulane University, New Orleans, Louisiana
  - Universidad de Cincinnati, Cincinnati, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sosa JA, Hanna JW, Robinson KA, Lanman RB. Increases in thyroid nodule fine-needle aspirations, operations, and diagnoses of thyroid cancer in the United States. Surgery. 2013 Dec;154(6):1420-6; discussion 1426-7. doi: 10.1016/j.surg.2013.07.006. Epub 2013 Oct 2. PMID 24094448
- [Background] Bongiovanni M, Spitale A, Faquin WC, Mazzucchelli L, Baloch ZW. The Bethesda System for Reporting Thyroid Cytopathology: a meta-analysis. Acta Cytol. 2012;56(4):333-9. doi: 10.1159/000339959. Epub 2012 Jul 25. PMID 22846422
- [Background] Hodak SP, Rosenthal DS; American Thyroid Association Clinical Affairs Committee. Information for clinicians: commercially available molecular diagnosis testing in the evaluation of thyroid nodule fine-needle aspiration specimens. Thyroid. 2013 Feb;23(2):131-4. doi: 10.1089/thy.2012.0320. Epub 2012 Nov 27. PMID 22984796
- [Background] Nikiforova MN, Wald AI, Roy S, Durso MB, Nikiforov YE. Targeted next-generation sequencing panel (ThyroSeq) for detection of mutations in thyroid cancer. J Clin Endocrinol Metab. 2013 Nov;98(11):E1852-60. doi: 10.1210/jc.2013-2292. Epub 2013 Aug 26. PMID 23979959
- [Background] Ali SZ, Fish SA, Lanman R, Randolph GW, Sosa JA. Use of the afirma(R) gene expression classifier for preoperative identification of benign thyroid nodules with indeterminate fine needle aspiration cytopathology. PLoS Curr. 2013 Feb 11;5:ecurrents.eogt.e557cbb5c7e4f66568ce582a373057e7. doi: 10.1371/currents.eogt.e557cbb5c7e4f66568ce582a373057e7. PMID 23437421